CLINICAL TRIAL: NCT02993003
Title: Optimal Positioning of Nasopharyngeal Temperature Probes in Pediatric Patients: A Prospective Cohort Study
Brief Title: Optimal Positioning of Nasopharyngeal Temperature Probes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No enrollment
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15-1216
Record Dates: First submitted 2016-07-18; First posted 2016-12-14 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Accuracy of Nasopharyngeal Probes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Children between 7 months and 12 months (Other): nasopharyngeal probe will be marked with indelible ink from 2-10 cm in 1-cm increments and inserted 10 cm
  Interventions: Device: Nasopharyngeal probe
- children between 1 and 5 years (Other): nasopharyngeal probe will be marked with indelible ink from 2-15 cm in 1.5-cm increments and inserted 10 cm
  Interventions: Device: Nasopharyngeal probe
- children between 6 and 12 years (Other): a nasopharyngeal probe will be marked with indelible ink from 2 to 20 cm at 2 cm increments from its tip, and inserted 20 cm
  Interventions: Device: Nasopharyngeal probe

INTERVENTIONS:
Device: Nasopharyngeal probe — nasopharyngeal probe insertion

SUMMARY:
Core temperature is of greatest interest in terms of temperature monitoring as it is thought to represent the temperature of the vessel-rich groups that are instrumental in thermoregulatory control. The nasopharynx is among the recommended temperature monitoring sites for core body temperature. It is the part of the pharynx that lies above the soft palate. Anteriorly it opens to the nasal cavities through the choanae; inferiorly it communicates with the oropharynx through the pharyngeal isthmus. Nasopharyngeal temperatures are accurate in adults when probes are inserted between 10 and 20 cm.

The optimal depth for insertion of nasopharyngeal probes remains poorly defined in infants and children. While some data suggest that anthropometric measurements are well correlated with endoscopic measurements in infants based on weight, the accuracy of temperature measurements at these and other distances has yet to be quantified. The investigators thus propose to determine the insertion depth (or range of depths) for nasopharyngeal temperature proves that best approximate core temperature as measured in the distal esophagus in infants and children of various sizes. The comparison site will be the distal esophagus since there is broad consensus that the distal third of the esophagus it at core-body temperature.

For the two groups of infants aged up to twelve months, the nasopharyngeal probe will be marked with indelible ink from 2-10 cm in 1-cm increments and inserted 10 cm. For the two groups of children between 1 and 5 years, the nasopharyngeal probe will be marked with indelible ink from 2-15 cm in 1.5-cm increments and inserted 10 cm. For older children, a nasopharyngeal probe will be marked with indelible ink from 2 to 20 cm at 2 cm increments from its tip, and inserted 20 cm.

Both nasopharyngeal and esophageal temperatures will initially be recorded 30 minutes after induction of anesthesia. Nasopharyngeal probes will then be withdrawn at the designated increment for each age group and will be equilibrated for 5 minutes before the temperature is recorded. Thereafter, the nasopharyngeal withdrawal sequence will be repeated. The number of measurement will depend on the initial depth of insertion, with measurements continuing until only 2 centimeters remain in the nostril.

ELIGIBILITY:
Inclusion Criteria:

1. Elective non-cardiac surgery in children to last at least 1.5 hours;
2. Supine position anticipated;
3. General endotracheal anesthesia.

Exclusion Criteria:

1. Nasopharyngeal disease (e.g. sinusitis), upper airway abnormalities, or planned oral or facial surgery;
2. History of genetic or congenital anomalies leading to facial dimorphism;
3. History of recent substantive epistaxis or suspected bleeding disorder;
4. Therapeutic-dose anti-coagulation;
5. Contraindication to esophageal temperature probe insertion (i.e., esophageal varices, congenital anomalies).

Ages: 7 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
nasopharyngeal and esophageal temperatures | up to 2 hrs during surgery
  nasopharyngeal and esophageal temperatures at each depth

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sessler, M.D., Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No